CLINICAL TRIAL: NCT01994941
Title: Genotype Guided Versus Conventional Approach in Selection of Oral P2Y12 Receptor Blocker in Chinese Patients Suffering From Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Stephen Lee, Prof. Stephen Lee, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 13-402
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Platelet Reactivity; P2Y12 Receptor Blocker; CYP2C19 Genotyping
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genotype guided group (Experimental): Patients are given standard doses of clopidogrel (either 300mg or 600mg according to clinical protocol). Blood will be drawn for rapid genetic testing (Verigene) and results will be expected in 2-4 hours. If patients are intermediate or poor clopidogrel metabolisers, loading dose of ticagrelor 180mg are given to enhance the antiplatelet response.
  Apart from the approach in guiding the use of P2Y12 receptor blocker, all patients will be treated according to usual clinical care including medications and coronary intervention. Blood will also be sent to standard laboratory for CYP2C19 genotyping using conventional polymerase chain reaction (PCR) method so as to confirm the accuracy of rapid genetic test. 24 hours after initial clopidogrel loading, blood will be taken to measure platelet reactivity by verifyNow P2Y12 assay (Accumetrics). In case glycoprotein IIbIIIa inhibitor (Integrilin) is used, verifyNow P2Y12 assay will be performed 48 hours after cessation of Integrilin.
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor
- Clinical guided group (Active Comparator): Patients are given standard doses of clopidogrel (either 300mg or 600mg according to clinical protocol).
  Apart from the approach in guiding the use of P2Y12 receptor blocker, all patients will be treated according to usual clinical care including medications and coronary intervention. Blood will also be sent to standard laboratory for CYP2C19 genotyping using conventional polymerase chain reaction (PCR) method so as to confirm the accuracy of rapid genetic test. 24 hours after initial clopidogrel loading, blood will be taken to measure platelet reactivity by verifyNow P2Y12 assay (Accumetrics) which is an FDA approved, point-of-care device using light-transmission based optical detection which measures platelet aggregation. In case glycoprotein IIbIIIa inhibitor (Integrilin) is used, verifyNow P2Y12 assay will be performed 48 hours after cessation of Integrilin.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — A platelet aggregation inhibitor. Also a P2Y12 Receptor Blocker of a drug class Thienopyridine.
  Increasing evidence has shown that clopidogrel has wide inter-individual variability in pharmacokinetic and pharmacodynamic actions which lead to suboptimal antiplatelet effect especially in Asian population.
  A standard loading dose of 300mg or 600mg(according to clinical protocol) will be given to patients.
  Other Names: Plavix
Drug: Ticagrelor — A platelet aggregation inhibitor.
  Though this agent has better anti-ischemic effects, it is associated with increased bleeding risk especially in Chinese patients whom are considered to be more prone to bleeding complications.
  A loading dose of 180mg will be used.
  Other Names: Brilinta
  Arms: Genotype guided group

SUMMARY:
This study aims to compare the outcome between genotype guided versus clinical guided approach in selection of oral P2Y12 receptor blocker in Chinese patients suffering from acute coronary syndrome.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) is a disease with high mortality, morbidity and economic burden. Usually, it is caused by ischemic heart disease and atherosclerotic plaque rupture in the coronary arteries causing platelet activation, aggregation and thrombus formation. For decades, antiplatelet agents are the cornerstones of management of ACS and dual antiplatelet therapy with aspirin and P2Y12 receptor blocker are standard of care for patients with ACS with or without percutaneous coronary intervention. However, increasing evidence has shown that clopidogrel, which is a type of thienopyridine, has wide inter-individual variability in pharmacokinetic and pharmacodynamic actions which lead to suboptimal antiplatelet effect especially in Asian population. Cytochrome P450 2C19 is an important enzyme for thienopyridine metabolism and genetic polymorphisms of CYP2C19 have been demonstrated to be associated with clopidogrel resistance and ischemic event post percutaneous coronary intervention (1-3). The prevalence of the LOF allele of CYP2C19 is higher in Chinese than in Caucasians (4) and it may lead to the higher degree of clopidogrel resistance in Chinese patients as documented in our previous study (5) and study from another Asian country (6)

In view of the potential limitations of clopidogrel in ACS treatment, American and European guidelines recommend use of newer P2Y12 blockers such as ticagrelor (7) for ACS patients. Though these agents have better anti-ischemic effect, they are associated with increased bleeding risk especially in Chinese patients whom are considered to be more prone to bleeding complications. As a result, local physicians are reluctant in using these potent antiplatelet agents despite their proven clinical efficacy in Caucasian studies. Evidence has shown the correlation between CYP2C19 genotype, platelet reactivity, clinical outcome and currently CYP2C19 genotype is an emerging target in the pharmacogenomic approach in guiding the use of antiplatelet agents. With the advent of rapid genotyping technologies (8), it is anticipated that the appropriate drug can be given to the appropriate patient.

Verigene (Nanosphere, Northbrook, IL) is an FDA approved microarray-based genotyping assay for the rapid detection of cytochrome P450 2C19 polymorphisms from whole blood using nanoparticle probes. It utilises whole blood for detection of single nucleotide polymorphism and the results will be available in 2-4 hours. With proper training and handling, the accuracy is expected to be >99%. (9, 10)

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or above
* Diagnosis of Acute Coronary Syndrome
* P2Y12 receptor blocker naïve and planning for a loading dose of P2Y12 receptor blocker

Exclusion Criteria:

* Chronic renal failure on dialysis or plan for dialysis within 1 year
* Serious hepatic disease
* Active bleeding disorder
* Contraindicated or allergic to Clopidogrel or ticagrelor
* History of intracranial bleeding
* Women who are pregnant or who are of childbearing potential who do not use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity 24 hours after initial loading of clopidogrel measured by verifyNow P2Y12 assay | 24 hours
  Platelet reactivity 24 hours after initial loading of clopidogrel measured by verifyNow P2Y12 assay
Platelet reactivity 1 month after initial loading of clopidogrel measured by verifyNow P2Y12 assay | 1 month
  Platelet reactivity 1 month after initial loading of clopidogrel measured by verifyNow P2Y12 assay

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hospital Authority, Hong Kong, Hong Kong

REFERENCES:
- [Background] Mega JL, Simon T, Collet JP, Anderson JL, Antman EM, Bliden K, Cannon CP, Danchin N, Giusti B, Gurbel P, Horne BD, Hulot JS, Kastrati A, Montalescot G, Neumann FJ, Shen L, Sibbing D, Steg PG, Trenk D, Wiviott SD, Sabatine MS. Reduced-function CYP2C19 genotype and risk of adverse clinical outcomes among patients treated with clopidogrel predominantly for PCI: a meta-analysis. JAMA. 2010 Oct 27;304(16):1821-30. doi: 10.1001/jama.2010.1543. PMID 20978260
- [Background] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Myrand SP, Sekiguchi K, Man MZ, Lin X, Tzeng RY, Teng CH, Hee B, Garrett M, Kikkawa H, Lin CY, Eddy SM, Dostalik J, Mount J, Azuma J, Fujio Y, Jang IJ, Shin SG, Bleavins MR, Williams JA, Paulauskis JD, Wilner KD. Pharmacokinetics/genotype associations for major cytochrome P450 enzymes in native and first- and third-generation Japanese populations: comparison with Korean, Chinese, and Caucasian populations. Clin Pharmacol Ther. 2008 Sep;84(3):347-61. doi: 10.1038/sj.clpt.6100482. Epub 2008 Mar 19. PMID 18231117
- [Background] Chan MY, Tan K, Tan HC, Huan PT, Li B, Phua QH, Lee HK, Lee CH, Low A, Becker RC, Ong WC, Richards MA, Salim A, Tai ES, Koay E. CYP2C19 and PON1 polymorphisms regulating clopidogrel bioactivation in Chinese, Malay and Indian subjects. Pharmacogenomics. 2012 Apr;13(5):533-42. doi: 10.2217/pgs.12.24. PMID 22462746
- [Background] Chae H, Kim M, Koh YS, Hwang BH, Kang MK, Kim Y, Park HI, Chang K. Feasibility of a microarray-based point-of-care CYP2C19 genotyping test for predicting clopidogrel on-treatment platelet reactivity. Biomed Res Int. 2013;2013:154073. doi: 10.1155/2013/154073. Epub 2013 Mar 28. PMID 23607088
- [Background] Buchan BW, Peterson JF, Cogbill CH, Anderson DK, Ledford JS, White MN, Quigley NB, Jannetto PJ, Ledeboer NA. Evaluation of a microarray-based genotyping assay for the rapid detection of cytochrome P450 2C19 *2 and *3 polymorphisms from whole blood using nanoparticle probes. Am J Clin Pathol. 2011 Oct;136(4):604-8. doi: 10.1309/AJCPCPU9Q2IRNYXC. PMID 21917683
- [Background] Bernlochner I, Mayer K, Morath T, Orban M, Schulz S, Schomig A, Braun S, Kastrati A, Sibbing D. Antiplatelet efficacy of prasugrel in patients with high on-clopidogrel treatment platelet reactivity and a history of coronary stenting. Thromb Haemost. 2013 Mar;109(3):517-24. doi: 10.1160/TH12-08-0552. Epub 2013 Jan 17. PMID 23328965
- [Derived] Tam CC, Kwok J, Wong A, Yung A, Shea C, Kong SL, Tang WH, Siu D, Chan R, Lee S. Genotyping-guided approach versus the conventional approach in selection of oral P2Y12 receptor blockers in Chinese patients suffering from acute coronary syndrome. J Int Med Res. 2017 Feb;45(1):134-146. doi: 10.1177/0300060516677190. Epub 2016 Dec 22. PMID 28222641